CLINICAL TRIAL: NCT00733681
Title: A Prospective, Non-comparative Study to Evaluate the Performance of the DePuy P.F.C. Sigma Rotating Platform TC3 Knee Prosthesis in Revision Knee Arthroplasty.
Brief Title: The Press Fit Condylar (P.F.C.) Sigma Rotating Platform (RP) TC3 Revision Knee in Revision Knee Arthroplasty
Acronym: TC3
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subjects were no longer able to remain compliant with follow-up intervals
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 02/14
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty, Replacement, Knee; Prosthesis Failure; Revision surgery
MeSH Terms: conditions — Osteoarthritis; Prosthesis Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PFC Sigma RP TC3 Revision Knee System (Experimental): Revision knee surgery with the PFC Sigma RP TC3 Revision Knee System (mobile bearing).
  Interventions: Device: PFC Sigma RP TC3 Revision knee system

INTERVENTIONS:
Device: PFC Sigma RP TC3 Revision knee system — Orthopaedic implant system for revision total knee replacement
  Other Names: Sigma RP TC3

SUMMARY:
The purpose of this study is to evaluate the long-term clinical and functional performance of the P.F.C. Sigma Rotating Platform TC3 knee system in revision knee surgery and to determine whether the implant design results in a longer-lasting knee replacement.

DETAILED DESCRIPTION:
Primary outcome: Implant survival at 5 years Secondary Outcomes:Evidence of clinical and functional outcome determined by the Knee Society Score, anterior knee pain (Patellar Score). Evidence of health related quality of life determined by WOMAC OA index. Patient satisfaction at 1 and 5 years. Radiographic analysis according to Knee society guidelines. Implant survival annually to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over the age of 21 years (and skeletally mature).
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects whose primary diagnosis includes non-inflammatory or inflammatory degenerative joint disease.
* Subjects who require revision of any previous knee arthroplasty.
* Subjects who, in the opinion of the Clinical Investigator, are considered to be suitable for treatment with the investigation device, according to the indications specified in the package insert leaflet.
* Subjects who require revision of the femoral and/or tibial components. (Both components must be replaced as part of the study.)

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study (including malignancy, severe osteoporosis or disabling musculoskeletal problems).
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last 60 days (excluding any primary knee replacement study).
* Subjects who are currently involved in any injury litigation claims.
* Subjects with global instability, deficient extensor mechanism or severe bone loss (eg. due to fracture or tumour resection).
* Subjects who have had their contralateral knee replaced within the previous 6-month period.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2004-03; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Implant survival | 5 years

SECONDARY OUTCOMES:
Clinical/functional outcome (Knee Society & Patellar Scores). Health-related QoL (WOMAC OA Index). Patient Satisfaction at 1 & 5 years (2 patient questions). Radiographic analysis (Knee Society guidelines). Annual implant survival to 15 years. | 6 months, 1, 2, 3, 5, 10 and 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter J James, FRCS, Principal Investigator — City Hospital, Nottingham
Locations (9):
- CHU, Amiens, France
- Germany (2):
  - Orthopaedische Universitaetsklinik, Heidelberg
  - Asklepios Klinik, Lindenlohe
- Geneva University Hospital, Geneva, Switzerland
- United Kingdom (5):
  - Princess Alexandra Hospital NHS Site, Harlow, Essex
  - City Hospital, Nottingham, Nottinghamshire
  - Western Infirmary, Glasgow
  - Leicester General Infirmary, Leicester
  - Robert Jones & Agnes Hunt Orthopaedic Hospital, Oswestry